CLINICAL TRIAL: NCT07048730
Title: Gynecological and Fertility Impact of Allogeneic Hematopoietic Stem Cell Transplantation for Acute Leukemia Diagnosed in Adulthood (GYNEGRAFT)
Brief Title: Gynecological Impact of Allogeneic Hematopoietic Stem Cell Transplantation in Adults
Acronym: GYNEGRAFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2025/022
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Leukemia
Keywords: Acute leukemia; Allogeneic hematopoietic stem cell transplantation; Premature ovarian failure; Vulvovaginal graft-versus-host disease; Assisted reproductive technologies
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire (Experimental): A standardized questionnaire was specifically developed for the study to explore:
  * Women's socio-demographic data
  * Data about their hematological disease (type of leukemia, conditioning protocol, relapses, graft-versus-host disease etc.)
  * Information received by patients prior to transplantation concerning gynecological complications
  * Symptoms, screening, diagnosis and treatment of the main gynecological complications
  * Patients fertility (spontaneous or after assisted reproductive treatments)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A standardized questionnaire was specifically developed for the study to explore:
  * Women's socio-demographic data
  * Data about their hematological disease (type of leukemia, conditioning protocol, relapses, graft-versus-host disease etc.)
  * Information received by patients prior to transplantation concerning gynecological complications
  * Symptoms, screening, diagnosis and treatment of the main gynecological complications
  * Patients fertility (spontaneous or after assisted reproductive treatments)

SUMMARY:
Gynecological impact and infertility are major issues for women after allogeneic hematopoietic stem cell transplantation.

The aim of the present study is to investigate the prevalence of gynecological complications after allogeneic hematopoietic stem cell transplantation for acute leukemia in adulthood. By conducting a single-center retrospective descriptive analysis, the prevalence, follow-up and treatment of gynecological complications -including premature ovarian failure, vulvovaginal graft-versus-host-disease, cervical pathology- will be analysed

DETAILED DESCRIPTION:
Recent advances in the treatment of acute leukemia, notably through allogeneic hematopoietic stem cell transplantation, have markedly improved survival rates. However, these therapies are associated with significant gonadotoxic and immunosuppressive effects that adversely impact gynecological and reproductive health- including premature ovarian failure (POF), vulvovaginal graft-versus-host-disease and cervical pathology related to human papillomavirus (HPV) infection. POF is a very frequent complication that induce hypoestrogenic symptoms and long-term side effects such as osteoporosis and cardiovascular disease. POF also induce infertility; spontaneous pregnancies after allogeneic hematopoietic stem cell transplantation are very rare. In most cases, pregnancies are obtained thanks to oocyte donation. In oncology, recent advances in fertility preservation offer promising prospects, including in emergency situations. Among these approaches, ovarian cortex cryopreservation can be proposed. However, this method remains limited in hematology due to the risk of reintroducing residual leukemic cells when cryopreserved tissue is reused, a challenge that is currently an area of research. In this context, a specialist fertility consultation prior to allograft is recommended.

Most studies concerning gynecological impact of acute leukemia focus on patients transplanted during childhood and data concerning women diagnosed in adulthood is limited. Comprehensive evaluation of gynecological and fertility impact in women treated in adulthood is thus essential

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with acute leukemia, who underwent allogeneic hematopoietic stem cell transplantation in adulthood (>18 years),
* Aged 20 to 45 at the time of evaluation,
* At least 2 years post-transplant.
* French-speaking patients, without comprehension disorders, and literate,
* No objection to participation.

Exclusion Criteria:

* Premature ovarian failure prior to management of haemopathy, post-transplant relapse,
* Patient under legal protection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Gynecological complication after transplantation | 2 years
  Percentage of women who experienced at least one gynecological complication (premature ovarian failure, vulvovaginal graft-versus-host-disease or cervical pathology related to human papillomavirus infection) 2 years after transplantation.

SECONDARY OUTCOMES:
Information on gynecological complications | 2 years
  Percentage of women who received information on gynecological complications and infertility before allogeneic hematopoietic stem cell transplantation
Pre-transplant fertility consultations | 2 years
  Percentage of pre-transplant fertility consultations
Gynecological follow-up | 2 years
  Percentage of women having gynecological follow-up every six month or every year 2 years after allogeneic hematopoietic stem cell transplantation
Cervical cancer screening | 2 years
  Percentage of women with regular cervical cancer screening 2 years after allogeneic hematopoietic stem cell transplantation
HPV vaccination | 2 years
  Percentage of women vaccinated against HPV post-transplant
Hormone replacement therapy | 2 years
  Percentage of women with hormone replacement therapy 2 years after allogeneic hematopoietic stem cell transplantation
Bone mineral density | 2 years
  Percentage of women who have had a bone mineral density evaluation 2 years after allogeneic hematopoietic stem cell transplantation
Spontaneous or assisted pregnancy | 2 years
  Prevalence of spontaneous or assisted pregnancy after allogeneic hematopoietic stem cell transplantation
Psychological disorders | 2 years
  Prevalence of psychological disorders related to infertility or gynecological complications after allogeneic hematopoietic stem cell transplantation.
Risk factors associated with the occurrence of gynecological complications | 2 years
  Identification of risk factors associated with the occurrence of gynecological complications (conditioning, graft-versus-host disease, age, comorbidities, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France